CLINICAL TRIAL: NCT01047735
Title: Randomized Trial to Compare Surgical and Medical Treatments for Type 2 Diabetes (Triabetes) - Alliance of Randomized Trials of Medicine vs. Metabolic Surgery in Type 2 Diabetes ARMMST2D)
Brief Title: The TRIABETES - ARMMS-T2D Study: A Randomized Trial to Compare Surgical and Medical Treatments for Type 2 Diabetes
Acronym: TRIABETES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Anita P. Courcoulas, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20060163; RC1DK086037 (NIH); R01DK095128-01 (NIH)
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
Keywords: 21+ years old; Address; Adult; Amputation; Area; Arm; Atheroscleroses; Atherosclerosis; Atherosclerotic; Cardiovascular Disease; Bariatrics; Behavior Conditioning Therapy; Behavior Modification; Behavior Therapy; Behavior Treatment; Behavior or Life Style Modifications; Behavioral; Behavioral Conditioning Therapy; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Beta Cell; Blindness; Blood Pressure, High; Blood Vessels; Body Composition; Body Weight decreased; Cancers; Cardiac infarction; Cardiovascular Diseases; Care, Health; Cause of Death; Cell Function; Cell Process; Cell physiology; Cellular Function; Cellular Physiology; Cellular Process; Cessation of life; Clinical; Clinical Trials Design; Communities; Conditioning Therapy; Controlled Clinical Trials, Randomized; Controlled Study; Country; D-Glucose; Death; Decision Making; Dextrose; Diabetes Mellitus; Diabetes Mellitus, Adult-Onset; Diabetes Mellitus, Ketosis-Resistant; Diabetes Mellitus, Non-Insulin-Dependent; Diabetes Mellitus, Noninsulin Dependent; Diabetes Mellitus, Slow-Onset; Diabetes Mellitus, Stable; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type II; Diet; Disease; Disease remission; Disorder; Drugs; Dysfunction; Effectiveness; Epidemic; Functional disorder; Future; Gastric Bypass; Glucose; Health; Healthcare; Hepatic Disorder; Human, Adult; Hypertension; INFLM; Incidence; Inflammation; Insulin Cell; Insulin Resistance; Insulin Secreting Cell; Intestinal; Intestines; Intravenous Glucose Tolerance; Intravenous Glucose Tolerance Test; Kidney Failure; Kidney Insufficiency; Learning; Life Style; Life Style Modification; Lifestyle; Link; Liver diseases; Longitudinal Studies; MODY; Malignant Neoplasms; Malignant Tumor; Maturity-Onset Diabetes Mellitus; Measures; Medical; Medication; Metabolic; Methods; Modification; Morbid Obesity; Morbidity; Morbidity - disease rate; Mortality; Mortality Vital Statistics; Myocardial Infarct; Myocardial Infarction; NAFLD; NASH; NIDDM; Non-Insulin Dependent Diabetes; Non-Insulin-Dependent Diabetes Mellitus; Non-alcoholic steatohepatitis; Obesity; Obesity, Morbid; Operation; Operative Procedures; Operative Surgical Procedures; Outcome; Outcome Measure; PROV; Participant; Patients; Pharmaceutic Preparations; Pharmaceutical Preparations; Physical activity; Physiopathology; Pilot Projects; Population; Procedures; Programs (PT); Programs [Publication Type]; Provider; Psychosocial Factor; Public Health; RMSN; Randomized; Randomized Controlled Clinical Trials; Randomized Controlled Trials; Remission; Renal Failure; Renal Insufficiency; Reporting; Resolution; Science; Severe obesity; Structure; Subcellular Process; Surgical; Surgical Interventions; Surgical Procedure; T2D; T2DM; Testing; Type 2 diabetes; Type II diabetes; United States; Upper arm; Vascular Hypertensive Disease; Vascular Hypertensive Disorder; Weight; Weight Loss; Weight Reduction; Work; adiposity; adult human (21+); adult onset diabetes; atheromatosis; atherosclerotic vascular disease; bariatric surgery; behavior intervention; behavioral intervention; blood glucose regulation; body weight loss; bowel; cardiac infarct; cardiovascular disorder; cardiovascular risk; cardiovascular risk factor; clinical practice; comparative effectiveness; coronary attack; coronary infarct; coronary infarction; corpulence; corpulency; corpulentia; design; designing; diabetes; diabetic patient; disease/disorder; drug/agent; effective therapy; effectiveness research; fitness; gastric banding; gastric bypass surgery; glucose control; glucose homeostasis; glucose metabolism; glucose regulation; heart attack; heart infarct; heart infarction; hepatopathy; hyperpiesia; hyperpiesis; hypertensive disease; implantable gastric stimulation banding; insulin resistant; interest; ketosis resistant diabetes; life style intervention; lifestyle intervention; liver disorder; long-term study; malignancy; maturity onset diabetes; moderate obesity; neoplasm/cancer; non-alcohol fatty liver; non-alcohol induced steatohepatitis; non-alcoholic fatty liver; non-alcoholic steato-hepatitis; nonalcohol fatty liver; nonalcoholic fatty liver; nonalcoholic steato-hepatitis; nonalcoholic steatohepatitis; obese; obese people; obese person; obese population; obesity surgery; obesity, extreme; pathophysiology; pilot study; programs; psychosocial; psychosocial variables; public health medicine (field); public health relevance; randomisation; randomization; randomized controlled study; randomized trial; randomly assigned; respiratory; response; stomach bypass; stomach stapling; surgery; trial comparing; vascular; weight loss intervention; weight loss surgery; wt-loss
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Atherosclerosis; Cardiovascular Diseases; Behavior; Blindness; Hypertension; Neoplasms; Myocardial Infarction; Death; Diabetes Mellitus; Disease; Digestive System Diseases; Inflammation; Insulin Resistance; Renal Insufficiency; Liver Diseases; Obesity, Morbid; Non-alcoholic Fatty Liver Disease; Motor Activity; Body Weight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (3):
- Roux-en-Y Gastric Bypass Surgery (Experimental): Roux-en-Y Gastric Bypass Surgery
  Interventions: Procedure: Roux-en-Y Gastric Bypass Surgery
- Laparoscopic Adjustable Gastric Banding (Experimental): Laparoscopic Adjustable Gastric Banding
  Interventions: Procedure: Laparoscopic Adjustable Gastric Banding
- Lifestyle/Behavioral Weight Loss (Experimental): Lifestyle Weight Loss Intervention
  Interventions: Behavioral: Lifestyle Weight Loss Intervention

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass Surgery — Participants assigned to the Roux-en-Y Gastric Bypass treatment group will undergo a surgical procedure that limit foods intake and causes nutrients malabsorption. The procedure is performed with small incisions or laparoscopically. A small stomach pouch is created, the size of an egg, and the small intestine is connected to the pouch. Some of the stomach and small intestine are consequently bypassed by this anatomic change. Those in this treatment group will begin a gradual diet post surgery and will take life long vitamin supplements.
  Arms: Roux-en-Y Gastric Bypass Surgery
Procedure: Laparoscopic Adjustable Gastric Banding — Those assigned to the Laparoscopic Adjustable Gastric Banding study group will undergo a surgical procedure where an adjustable silicone band is placed around the upper stomach to decrease its capacity so that you will feel full sooner. It will assist in weight loss by helping you to limit intake of calories. The band will be placed by using several small incisions and telescopic instruments. A thin tube connects the band to an access port just under the skin that you may be able to feel but you will not be able to see it. This allows the band to be tightened or loosened to decrease or increase your stomach capacity as needed. The surgery will take on average 30-45 minutes.
  Other Names: LapBand
  Arms: Laparoscopic Adjustable Gastric Banding
Behavioral: Lifestyle Weight Loss Intervention — Participants will receive a standard behavior weight control program in an in-person format over a period of 12 months conducted by an experienced team of weight loss counselors. During the initial 6 months of study treatment, will attend weekly in-person individual sessions with a weight loss counselor. During months 7-12, will attend in-person sessions on the 1st and 3rd week of the month and will receive a brief (less than 10 minutes in duration) telephone call on the 2nd and 4th week of the month. Each session will focus on a specific behavioral topic related to weight loss, eating behaviors, or exercise behaviors.
  Arms: Lifestyle/Behavioral Weight Loss

SUMMARY:
This research study is being performed to begin to determine the effectiveness of two dominant bariatric surgery procedures versus an intensive lifestyle intervention to induce weight loss in patients and promote improvements in Type 2 diabetes mellitus (T2DM) in moderately obese patients.

T2DM is currently the 6th leading cause of mortality in the United States and is a major cause of kidney failure, blindness, amputations, heart attack, and other vascular and gastro-intestinal dysfunctions. Traditionally, treatments include intensive lifestyle modifications with or without glucose lowering agents. Neither treatment alone, or in combination, results in complete resolution of diabetes and its potential long-term complications. Bariatric surgery has been proven as an effective treatment to accomplish sustained and significant weight loss for those with severe obesity and has been shown to induce long-term remission of T2DM. However, despite enthusiasm for these potential treatment options, it is not clear whether diabetes is influenced by the type of surgery or by the amount of weight lost or if bariatric surgery is more effective than non-surgical weight loss induced by diet and physical activity in T2DM patients with moderate BMIs (30-40kg/m2; Class I and Class II obesity, or approximately 65-95 pounds overweight depending on your height). More well-controlled studies are needed to more completely inform health care decision making and clinical practice in this area. This research study aims to obtain preliminary information regarding the effectiveness of two major types of bariatric surgery, Laparoscopic Roux-en-Y Gastric Bypass and Laparoscopic Adjustable Gastric Banding versus an intensive lifestyle intervention to induce weight loss with diet and increased physical activity.

DETAILED DESCRIPTION:
The Specific Aims of the first phase of the study are as follows:

Aim 1. To determine the feasibility of performing a randomized trial comparing two major types of bariatric surgery, Laparoscopic Roux en Y Gastric Bypass (RNY) and Laparoscopic Adjustable Gastric Banding (GB) versus a lifestyle weight loss intervention (LWLI) induced by diet and increased physical activity in moderately obese patients (Class I and II obesity) with T2DM. We hypothesize that: 1) A randomized design with both surgical and non-surgical arms will be both feasible and acceptable to participants and to providers 2) There will be no difference in retention rates between the LWLI and surgical arms (RNY, GB) of the study and it will provide estimates of overall retention for future studies.

Aim 2. To obtain preliminary information regarding the effectiveness of two dominant bariatric surgery procedures versus an intensive lifestyle intervention to induce weight loss with diet and increased physical activity. We hypothesize that: 1) RNY will be superior to GB and LWLI in weight lost in 12 months.

Aim 3. To explore the feasibility, methods for, and implementation of a range of early outcome measures including; resolution of diabetes, glucose control, medication usage, insulin resistance, beta cell function, body composition, objective measures of physical activity, and several psychosocial measures. We hypothesize that: 1) Participants will be willing to undergo a range of early outcome testing measures to assess metabolic change, body composition alterations, objective physical activity, and psychosocial factors. 2) Measures of T2DM improvement including an intravenous glucose tolerance test (IVGTT) will be feasible in a subset of participants in each study arm and RNY will be superior to both GB and LWLI for the clinical and metabolic improvement of T2DM. 3) The LWLI group will show improvements in physical activity compared to RNY and GB.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 55 years
* Mild to moderate obesity with a BMI between 30 and 40 kg/m2
* For potential subjects with BMI 35 to 40 kg/m2: T2DM confirmed by either a documented fasting blood glucose > 126 mg/dl OR treatment with an anti-diabetic medication
* For potential subjects with BMI 30 to 35 kg/m2: T2DM that is difficult to control medically and is recommended for the study by the subject's endocrinologist AND treatment with an anti-diabetic medication
* Willingness to be randomized to a surgical intervention

Exclusion Criteria:

* Prior bariatric or foregut surgery
* Poor overall general health
* Impaired mental status
* Drug and/or alcohol addiction
* Current smoking
* Pregnant or plans to become pregnant
* Type 1 Diabetes Mellitus
* Portal hypertension and/or Cirrhosis
* Failed study-related nutrition or psychological assessment
* Current participation in any other research study
* Inability to provide informed consent
* Unlikely to comply with study protocol
* Unable to communicate with study staff
* Unable to exercise (walk a city block or a flight of stairs)

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of performing a randomized trial comparing two major types of bariatric surgery versus a lifestyle weight loss intervention (LWLI) induced by diet and increased physical activity in moderately obese patients with T2DM. | 6 months, 1 year

SECONDARY OUTCOMES:
Preliminary information regarding the effectiveness of two dominant bariatric surgery procedures versus an intensive lifestyle intervention to induce weight loss with diet and increased physical activity. | 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anita P Courcoulas, MD, MPH, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- William F Gourash, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Courcoulas AP, Goodpaster BH, Eagleton JK, Belle SH, Kalarchian MA, Lang W, Toledo FG, Jakicic JM. Surgical vs medical treatments for type 2 diabetes mellitus: a randomized clinical trial. JAMA Surg. 2014 Jul;149(7):707-15. doi: 10.1001/jamasurg.2014.467. PMID 24899268
- [Background] Courcoulas AP, Gallagher JW, Neiberg RH, Eagleton EB, DeLany JP, Lang W, Punchai S, Gourash W, Jakicic JM. Bariatric Surgery vs Lifestyle Intervention for Diabetes Treatment: 5-Year Outcomes From a Randomized Trial. J Clin Endocrinol Metab. 2020 Mar 1;105(3):866-76. doi: 10.1210/clinem/dgaa006. PMID 31917447
- [Background] Courcoulas AP, Belle SH, Neiberg RH, Pierson SK, Eagleton JK, Kalarchian MA, DeLany JP, Lang W, Jakicic JM. Three-Year Outcomes of Bariatric Surgery vs Lifestyle Intervention for Type 2 Diabetes Mellitus Treatment: A Randomized Clinical Trial. JAMA Surg. 2015 Oct;150(10):931-40. doi: 10.1001/jamasurg.2015.1534. PMID 26132586